CLINICAL TRIAL: NCT02201862
Title: Non-Invasive Chromosomal Evaluation of Trisomy Study
Acronym: NICHE
Status: Completed | Type: Observational
Sponsor: Cindy Cisneros (Industry)
Responsible Party: Sponsor-Investigator, Cindy Cisneros, CRA, Roche Sequencing Solutions
Organization: Roche Sequencing Solutions (Industry)
Other Study IDs: AD201
Record Dates: First submitted 2014-07-22; First posted 2014-07-28 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Aneuploidy; Trisomy 21; Trisomy 18; Trisomy 13; Down Syndrome
Keywords: Aneuploidy; Down Syndrome; amniocentesis; chronic villus sampling; Trisomy; non-invasive prenatal testing; Chromosome disorders
MeSH Terms: conditions — Aneuploidy; Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Trisomy; Chromosome Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Euploid Subjects: Subject's with fetal euploidy confirmed by chromosome analysis
- Aneuploid Subjects: Subject's with fetal aneuploidy confirmed by chromosome analysis

SUMMARY:
This study is being conducted to provide clinically annotated samples to support continued improvements in the Ariosa Test content, methodology, specimen processing and quality control.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is at least 18 years old and can provide informed consent;
* 2. Subject has a viable singleton or twin pregnancy;
* 3. Subject is confirmed to be at least 10 weeks, 0 days gestation at the time of the study blood draw;
* 4. Subject is planning to undergo CVS and/or amniocentesis for the purpose of genetic analysis of the fetus OR the subject has already undergone CVS and/or amniocentesis and is known to have a fetus with a chromosomal abnormality confirmed by genetic analysis.

Exclusion Criteria:

* 1. Subject has known aneuploidy;
* 2. Subject is pregnant with more than two fetuses or has had sonographic evidence of three or more gestational sacs at any time during pregnancy;
* 3. Subject has a fetal demise (including natural or elective reduction) identified prior to consent;
* 4. Subject has history of malignancy treated with chemotherapy and/or major surgery, or bone marrow transplant;

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women planning to undergo chorionic villus sampling (CVS) and/or amniocentesis for the purpose of genetic evaluation of the fetus.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Detection of aneuploidy | 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University California San Diego, San Diego, California
  - Women's Healthcare Group of PA, Oaks, Pennsylvania
  - Regional Obestrical Consultants, Chattanooga, Tennessee

REFERENCES:
- [Background] Norton ME, Brar H, Weiss J, Karimi A, Laurent LC, Caughey AB, Rodriguez MH, Williams J 3rd, Mitchell ME, Adair CD, Lee H, Jacobsson B, Tomlinson MW, Oepkes D, Hollemon D, Sparks AB, Oliphant A, Song K. Non-Invasive Chromosomal Evaluation (NICE) Study: results of a multicenter prospective cohort study for detection of fetal trisomy 21 and trisomy 18. Am J Obstet Gynecol. 2012 Aug;207(2):137.e1-8. doi: 10.1016/j.ajog.2012.05.021. Epub 2012 Jun 1. PMID 22742782